CLINICAL TRIAL: NCT00004493
Title: Phase II Pilot Randomized Study of Sodium Dichloroacetate in Patients With Congenital Lactic Acidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/14274; UCSD-FDR001481
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-05

CONDITIONS: Lactic Acidosis
Keywords: inborn errors of metabolism; lactic acidosis; rare disease
MeSH Terms: conditions — Acidosis, Lactic; Metabolism, Inborn Errors; Rare Diseases | interventions — Dichloroacetic Acid

INTERVENTIONS:
Drug: sodium dichloroacetate

SUMMARY:
OBJECTIVES: I. Determine the pharmacokinetics of sodium dichloroacetate (DCA) in patients with congenital lactic acidemia.

II. Determine the efficacy of DCA in decreasing the frequency and/or severity of acute episodes of acidotic illness, improving linear growth, improving neurological or developmental function, or slowing neurological or developmental deterioration in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, cross over study. Patients are randomized to start with one of two different doses of sodium dichloroacetate (DCA).

Patients receive one of two doses of oral DCA for 6 months, then switch to the alternate dose for 6 months. This course is repeated once.

Patients are followed for up to 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of stable, persistent lactic acidemia Venous lactate at least 3 mM under basal conditions defined as: At least 4 hours postprandial No concurrent illness

OR

* Diagnosis of cerebral lactic acidemia with elevated lactic acid in CSF but not in the blood
* No organic acidemias or defective gluconeogenesis

--Patient Characteristics--

* Hematopoietic: Hemoglobin at least 7 mg/dL
* Hepatic: Bilirubin no greater than 3 times upper limit of normal (ULN) AST, ALT, or GGT no greater than 10 times ULN
* Renal: Creatinine no greater than 2 mg/dL
* Cardiovascular: Ejection fraction at least 25%
* Other: No hypoglycemia (blood sugar less than 50 mg/dL at no greater than 12 hours fasting) No severe peripheral neuropathy interfering with normal activities of living

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 1998-09; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barshop, Study Chair — University of California, San Diego
Locations (1):
- University of California San Diego School of Medicine, La Jolla, California, United States